CLINICAL TRIAL: NCT02986555
Title: Virtual Reality Stress and Relief Project, Research on Quantification of VR Related Stress, Motion Sickness and Visual Fatigue
Brief Title: Research on Quantification of VR(Virtual Reality) Related Stress and Relaxation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Samsung Electronics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2016-10-007
Record Dates: First submitted 2016-12-02; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Stress, Psychological; Motion Sickness; Visual Fatigue
Keywords: Stress; Virtual Reality; Motion sickness; Visual Fatigue; Biofeedback
MeSH Terms: conditions — Stress, Psychological; Motion Sickness; Asthenopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stress relief with existing biofeedback (Placebo Comparator): After distressing virtual reality video and full resting time to relieve this stress, the investigators are going to give cognitive distress with serial seven, accompanied with existing biofeedback approach to relieve stress.
  Interventions: Device: Existing Biofeedback
- Stress relief with biofeedback and VR (Active Comparator): After distressing virtual reality video and full resting time to relieve this stress, the investigators are going to give cognitive distress with serial seven, accompanied with biofeedback combined to virtual reality relaxation.
  Interventions: Device: Biofeedback accompanied with virtual reality

INTERVENTIONS:
Device: Existing Biofeedback — Using relaxing assisted biofeedback approach
  Arms: Stress relief with existing biofeedback
Device: Biofeedback accompanied with virtual reality — Using relaxation approach with existing biofeedback accompanied by virtual reality relaxation
  Arms: Stress relief with biofeedback and VR

SUMMARY:
Current virtual reality device makes motion sickness and visual fatigue having limitation for recreation and other clinical approaches. Still there is no standardized quantification of motion sickness and visual fatigue measurement with objective approach. Current biofeedback accompanied with virtual reality would be promising tool for stress relief.

DETAILED DESCRIPTION:
Current virtual reality device makes motion sickness and visual fatigue having limitation for recreation and other clinical approaches. Still there is no standardized quantification of motion sickness and visual fatigue measurement with objective approach. After quantification and improvement with these shortcomings, current biofeedback accompanied with virtual reality would be promising tool for stress relief. This research aims to measure objective motion sickness and visual fatigue with psychological stress in highly stressed group, and to compare between stress relief with existing biofeedback only approach and relief with mixed biofeedback and virtual reality relaxation.

ELIGIBILITY:
Inclusion Criteria:

* scored at least 20 on the PSS-10 (Perceived Stress Scale 10) to verify highly psychological stressed participants at the baseline visits.

Exclusion Criteria:

* the existence of a current Major depressive disorder or panic disorder, psychotic disorder (e.g., schizophrenia or delusional disorder), bipolar affective disorder,active alcohol or drug use disorder, neurological illness including significant cognitive impairment or Parkinson's disease, mental retardation, significant medical conditions, epilepsy, histories of alcohol or drug dependence, personality disorders, or brain damages during the screening and baseline visits, per the Mini-International Neuropsychiatric Interview (Sheehan et al., 1998) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5)
* the existence of active disease in both orbital parts

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Change of Heart rate variability especially ratio of High Frequency and Low Frequency | Baseline, after 64minutes and 30 seconds (which means cognitive distress stimuli,Serial Seven), after 85 minutes 30 seconds (after completing biofeedback or biofeedback with virtual reality relaxation)

SECONDARY OUTCOMES:
Change of Respiration Rate | Baseline, after 64minutes and 30 seconds (which means cognitive distress stimuli,Serial Seven), after 85 minutes 30 seconds (after completing biofeedback or biofeedback with virtual reality relaxation)
Psychological distress scale with Perceived Stress Scale 10 | Baseline, after 64minutes and 30 seconds (which means cognitive distress stimuli,Serial Seven), after 85 minutes 30 seconds (after completing biofeedback or biofeedback with virtual reality relaxation)
Visual analogue scale for motion sickness | Baseline, after 64minutes and 30 seconds (which means cognitive distress stimuli,Serial Seven), after 85 minutes 30 seconds (after completing biofeedback or biofeedback with virtual reality relaxation)
Visual analogue scale for negative emotion | Baseline, after 64minutes and 30 seconds (which means cognitive distress stimuli,Serial Seven), after 85 minutes 30 seconds (after completing biofeedback or biofeedback with virtual reality relaxation)
Visual analogue scale for visual fatigue | Baseline, after 64minutes and 30 seconds (which means cognitive distress stimuli,Serial Seven), after 85 minutes 30 seconds (after completing biofeedback or biofeedback with virtual reality relaxation)

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jin Jeon, M.D.,Ph.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, Irwon-dong, Gangnam-gu, South Korea

IPD SHARING:
Plan to Share IPD: No